CLINICAL TRIAL: NCT05395871
Title: Investigating the Use of Behavioural Science Informed Messages to Facilitate Attendance at Breast Cancer Screening
Brief Title: Behavioural Science Messages in Breast Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: NHS England (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 22IC7498
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Results first posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer Screening; Behavioural Science; Mobile Messaging; Behavioural Interventions; Healthcare Inequalities
MeSH Terms: conditions — Breast Neoplasms | interventions — Videotape Recording

STUDY DESIGN:
Intervention Model Description: 3 arm randomised controlled trial
Who Masked: Care Provider
Masking Description: The screening services will not have access to the allocation of participants and will be masked. They will not be able to determine which messages are being sent to different women being invited to screen, as allocation will be undertaken by the third party messaging company following provision of a screening invitation list by the service.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (Active Comparator): A text message sent 7 days prior then 48 hours before a booked/timed appointment. The content of the message will be the 'usual care' content that is currently sent by the London Breast Cancer Screening Programme. This includes a link to a YouTube hosted video.
  Interventions: Other: Usual Care Message
- Behavioural Message (Experimental): A text message sent 7 days prior then 48 hours before a booked/timed appointment. The content of the message has been informed by previous co-design work, and incorporate behavioural change techniques. This will include the same link to a YouTube hosted video, as the usual care arm.
  Interventions: Behavioral: Behavioural Message
- Behavioural Message + Video (Experimental): An text message sent 7 days prior then 48 hours before a booked/timed appointment. The content of the message will be the same as the Behavioural text, however the link will be replaced with a weblink to an animated video. This video has been designed through an extensive co-design process involving several behavioural change techniques designed to overcome barriers highlighted in this qualitative work.
  Interventions: Behavioral: Behavioural Message + Video

INTERVENTIONS:
Behavioral: Behavioural Message — Messaging involving increased salience, increasing positive emotions and information on health consequences
  Arms: Behavioural Message
Behavioral: Behavioural Message + Video — Messaging as above. The video also includes information on emotional consequences, problem solving, anticipated regret, reducing negative emotions and credible source techniques.
  Arms: Behavioural Message + Video
Other: Usual Care Message — Standard usual care message involving link to non-behavioural science informed video
  Arms: Usual Care

SUMMARY:
Breast cancer is the most common cancer in the United Kingdom, with 1 in 8 women affected during their lifetime. Whilst survival rates are high, the 5-year survival rate is 72% higher with the earliest stage breast cancer, compared to the latest disease stage. The National Health Service Breast Screening Programme invites women aged 50 to 70 years old every three years to a mammogram. By enabling earlier detection, it is estimated that the National Health Service Breast Screening Programme saves 1300 lives per year.

Despite the potential benefits of breast cancer screening, attendance is falling. Behavioural Science is a field of study concerning understanding the processes underpinning human action. Behavioural theories, such as the Capability Opportunity Motivation-Behaviour model. Recent studies have shown the application of behavioural science to screening may also facilitate uptake of invitations. However, the use of plain text messages limits which behavioural determinants can be feasibly addressed, and what techniques can be used. Video messages can allow for more complex and a broader range of behavioural change techniques to be incorporated, and therefore have greater impact upon attendance.

Whilst behavioural science-informed messages have previously been trialed by groups to facilitate breast screening attendance, their effectiveness has been variable. One of the reasons for this, is that text messages are of limited length and formatting capability, thus restricting the number of behavioural change techniques that can be included. Moreover, some behavioural techniques are more complex than others, and plain text can limit the extent to which these can be feasibly incorporated. Video messaging provides a delivery mechanism that may enable more complex, and different combinations to be trialed. There is however, a paucity of data regarding the impact of sending a video-based behavioural science message upon attendance rates at breast cancer screening programmes. This study looks to investigate the impact of a video-message, compared to behavioural science-based text messages and standard reminder messages.

The primary object is to determine the impact of behavioural science informed (1) video and (2) text messages compared to usual care, upon uptake of breast cancer screening. Secondary objectives involve how this impact on attendance differs between population subgroups including people from differing demographic groups.

DETAILED DESCRIPTION:
This study will be conducted as a randomised control trial in the London screening region of the National Health Service Breast Screening Programme. The study will last over 6 months. The administrative hub for the National Health Service Breast Screening Programme. in London is based at the Royal Free Hospital, who will oversee invitation scheduling, message delivery and outcome data collation through their existing delivery systems.

Participants will be randomised using simple randomisation method in a 1:1:1 fashion to either intervention arm or usual care. Randomisation will utilise a computerised system in which each participant who is due for screening in the study period is randomly allocated a number corresponding to the message they will receive. This will be undertaken by the screening hub, and will be passed on to the message delivery service who will ensure the correct template is sent.

Written invitations are sent, as standard practice, by the National Health Service Breast Screening Programme. to invite women to either (1) an appointment at a set time, date and location (so-called timed invitations) or (2) to call and book an appointment (or open invitation). Following this, as part of usual care, those selected for open invitations will receive a first text message 7 days post written invitation. They will then receive two text message reminders, 7 days and 2 days prior to the appointment, once it has been booked. Those who receive timed invitations will just receive the two reminder messages, 7 and 2 days prior to the appointment. The decision to offer an individual a timed or open invitation is made by the screening service based on their pandemic recovery process, and will not be altered by this project.

This randomised controlled trial will involve randomising participants to receive the usual care messages (according to the timings outlined above), a plain text message incorporating or the behavioural message with a new link to a video incorporating more behavioural techniques.

The content of the intervention messages, and the video have been developed through extensive Patient and Public Involvement and Engagement work including 10 interviews, 2 focus groups and 2 co-design workshops. Members of the public have been consulted throughout the process, especially regarding the representations of individuals in the video, and the message content. The feedback received has been used to alter the materials, and further feedback received. Through this iterative approach we have ensured content is appropriate. We have also sought feedback from members of community groups working in mental health services specifically for African Caribbean and Arabic Speaking adults, and trans-led organisation to improve the quality of life of trans people, to ensure individuals from these groups are happy with representations. Screening commissioners at National Health Service England have also approved this content. The National Health Service Identity team have provided approvals for the use of National Health Service logos/branding, and the team at London Northwest Healthcare National Health Service Trust approved the use of their name.

The video will be hosted on a private page on the Imperial College London website, which will be available only to those who have been sent the link. The video will be translated into several languages, with voice overs also available in different languages, to ensure people from a diverse background are able to understand the content.

After 3 months from the initial written invitations, data will be collated from the breast screening hub regarding whether an individual attended an appointment and whether the messages were successfully sent. This will be repeated at 6 months corresponding to the key performance indicator of the service.

ELIGIBILITY:
The inclusion criteria will match those used by the National Health Service Breast Screening Programme, as all invitations will come directly from the programme, as per usual care. These include:

* Aged between 50 to 70 at the time of invitation
* Lives within London screening region
* Registered as female with primary care physician

The exclusion criteria will match those used by the National Health Service Breast Screening Programme, as all invitations will come directly from the programme, as per usual care. These include:

* Previous attendance at breast screening in the current (3-year cycle)
* Opted out of receiving text messages
* Opted out of screening
* Previous bilateral mastectomy

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Registered with primary care physician as female and therefore will be invited to the breast cancer screening programme
Enrollment: 34047 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ara Darzi, FRCS, Principal Investigator — Imperial College London
Locations (1):
- NHS Breast Screening Hub, Edgware, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kerrison RS, Shukla H, Cunningham D, Oyebode O, Friedman E. Text-message reminders increase uptake of routine breast screening appointments: a randomised controlled trial in a hard-to-reach population. Br J Cancer. 2015 Mar 17;112(6):1005-10. doi: 10.1038/bjc.2015.36. PMID 25668008
- [Background] Acharya A, Sounderajah V, Ashrafian H, Darzi A, Judah G. A systematic review of interventions to improve breast cancer screening health behaviours. Prev Med. 2021 Dec;153:106828. doi: 10.1016/j.ypmed.2021.106828. Epub 2021 Oct 5. PMID 34624390
- [Background] Michie S, van Stralen MM, West R. The behaviour change wheel: a new method for characterising and designing behaviour change interventions. Implement Sci. 2011 Apr 23;6:42. doi: 10.1186/1748-5908-6-42. PMID 21513547
- [Background] NHS Digital. Breast Screening Programme, England 2019-20 [Internet]. 2021 [cited 2021 Jun 14]. Available from: https://digital.nhs.uk/data-and-information/publications/statistical/breast-screening-programme/england---2019-20
- [Background] Huf S, Kerrison RS, King D, Chadborn T, Richmond A, Cunningham D, Friedman E, Shukla H, Tseng FM, Judah G, Darzi A, Vlaev I. Behavioral economics informed message content in text message reminders to improve cervical screening participation: Two pragmatic randomized controlled trials. Prev Med. 2020 Oct;139:106170. doi: 10.1016/j.ypmed.2020.106170. Epub 2020 Jun 29. PMID 32610059
- [Derived] Acharya A, Darzi A, Judah G. An SMS and animated video intervention to increase uptake of breast cancer screening: a randomised controlled trial. Lancet. 2023 Nov;402 Suppl 1:S17. doi: 10.1016/S0140-6736(23)02133-5. PMID 37997056
- [Derived] Acharya A, Ashrafian H, Cunningham D, Ruwende J, Darzi A, Judah G. Evaluating the impact of a novel behavioural science informed animation upon breast cancer screening uptake: protocol for a randomised controlled trial. BMC Public Health. 2022 Jul 19;22(1):1388. doi: 10.1186/s12889-022-13781-x. PMID 35854267

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | Behavioural Message | Behavioural Message + Video
Started | 11748 (Combined Open and Timed Appointments) | 11047 (Combined Open and Timed Appointments) | 11252 (Combined Open and Timed Appointments)
Completed | 11748 | 11047 | 11252
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Behavioural Message | Behavioural Message + Video | Total
Number analyzed (Participants) | 11748 | 11047 | 11252 | 34047
Age, Customized [Median (Inter-Quartile Range); unit: years] — The ranges demonstrated are inter-quartile ranges, not full ranges thus the age for the lower quartile for the usual care group is lower than for the total group. Population: Note of the overall population equals to 34047 participants.
  Total = Timed (9027) + Open (25020) = 34047
  Usual care = 3094 + 8654 = 11748 Behavioural message = 2952 + 8095 = 11047 Behavioural mesage + Video = 2981 + 8271 = 11252
  9027 received timed invitaitons (3094 usual care, 2952 Behavioural Message and 2981 Behavioural Message + Video). 25020 received open invitations (8654 usual care, 8095 Behavioural Message and 8271 Behavioural Message + Video)
  years
    Timed: number analyzed (Participants) | 3094 | 2952 | 2981 | 9027
    Timed | 59 [53 to 64] | 59 [54 to 64] | 59 [54 to 64] | 59 [54 to 64]
    Open: number analyzed (Participants) | 8654 | 8095 | 8271 | 25020
    Open | 58 [52 to 63] | 58 [53 to 63] | 57 [52 to 63] | 58 [52 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11748 | 11047 | 11252 | 34047
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White | 4000 | 3804 | 3818 | 11622
  Ethnicity: Black | 810 | 758 | 786 | 2354
  Ethnicity: Asian | 1401 | 1328 | 1359 | 4088
  Ethnicity: Mixed | 133 | 126 | 132 | 391
  Ethnicity: Other | 360 | 312 | 335 | 1007
  Ethnicity: Not stated | 5044 | 4719 | 4822 | 14585
Region of Enrollment [Number; unit: participants]
  United Kingdom | 11748 | 11047 | 11252 | 34047
IMD Decile [Count of Participants; unit: Participants] — IMD denotes the Index of Multiple Deprivation. Pre-defined areas (called LSOAs) of the UK are ranked from the most deprived area to the least deprived area. The deciles represent the least deprived (IMD 10) 10% of areas to the most deprived 10% of areas (IMD 1).
  Numbers represent the no. of participants living in these areas within the study groups.
  Participants
    IMD 1 | 160 | 175 | 214 | 549
    IMD 2 | 1108 | 992 | 1008 | 3108
    IMD 3 | 1335 | 1164 | 1344 | 3843
    IMD 4 | 1512 | 1455 | 1438 | 4405
    IMD 5 | 1465 | 1436 | 1383 | 4284
    IMD 6 | 1555 | 1519 | 1511 | 4585
    IMD 7 | 1446 | 1312 | 1302 | 4060
    IMD 8 | 1383 | 1291 | 1318 | 3992
    IMD 9 | 1136 | 1118 | 1151 | 3405
    IMD 10 | 625 | 557 | 550 | 1732
    Not stated | 23 | 28 | 33 | 84
Invitation Type (open/timed) [Count of Participants; unit: Participants]
  Timed | 3094 | 2952 | 2981 | 9027
  Open | 8654 | 8095 | 8271 | 25020

OUTCOME MEASURES:

1. Primary Outcome: No. of Participants Taking up Breast Cancer Screening at Three Months- Intention to Treat
Description: Percentage uptake of breast cancer screening, three months after the initial invitation letter- intention to treat.
Time Frame: 3 months
Population: Timed invitation
Measure: Number; unit: participants
Arm/Group | Usual Care | Behavioural Message | Behavioural Message + Video
Number analyzed (Participants) | 3094 | 2952 | 2981
participants | 2225 | 2064 | 2137

2. Primary Outcome: No. of Participants Taking up Breast Cancer Screening at Three Months- Per Protocol
Description: No. of participants taking up breast cancer screening, three months after the initial invitation letter- per protocol
Time Frame: 3 months
Population: Timed Appointments
Measure: Number; unit: participants
Arm/Group | Usual Care | Behavioural Message | Behavioural Message + Video
Number analyzed (Participants) | 2721 | 2535 | 2615
participants | 2073 | 1899 | 1977

3. Secondary Outcome: No. of Participants Taking up Breast Cancer Screening, Three Months After the Initial Invitation Amongst Those From Sociodemographic Groups (Deprivation, Ethnicity)
Description: No. of participants taking up breast cancer screening, three months after the initial invitation letter amongst those from sociodemographic groups (ethnicity)
  Note there remain 3 trial arms (usual care, behavioural message, behavioural message + video), data represents subgroup analysis dichotomising these arms into white v. non white ethnicity).
Time Frame: 3 months
Population: Timed appointments
Measure: Number; unit: participants
Arm/Group | Usual Care | Behavioural Message | Behavioural Message + Video
Number analyzed (Participants) | 3094 | 2952 | 2981
participants
  White: number analyzed (Participants) | 1596 | 1473 | 1501
  White | 1379 | 1276 | 1303
  Non- White: number analyzed (Participants) | 1498 | 1479 | 1480
  Non- White | 1206 | 1194 | 1243

4. Secondary Outcome: No. of Participants Taking up Uptake of Breast Cancer Screening, Three Months After the Initial Invitation Letter, Amongst Those Given Different Invitation Types.
Description: No. of participants taking up breast cancer screening, three months after the initial invitation letter, amongst those given different invitation types.
Time Frame: 3 months
Population: Open Invitations
Measure: Number; unit: participants
Groups:
- Usual Care- Open: A text message sent 7 days prior then 48 hours before a booked/timed appointment. The content of the message will be the 'usual care' content that is currently sent by the London Breast Cancer Screening Programme. This includes a link to a YouTube hosted video.
  Usual Care Message: Standard usual care message involving link to non-behavioural science informed video
- Behavioural Message- Open: A text message sent 7 days prior then 48 hours before a booked/timed appointment. The content of the message has been informed by previous co-design work, and incorporate behavioural change techniques. This will include the same link to a YouTube hosted video, as the usual care arm.
  Behavioural Message: Messaging involving increased salience, increasing positive emotions and information on health consequences
- Behavioural Message + Video- Open: An text message sent 7 days prior then 48 hours before a booked/timed appointment. The content of the message will be the same as the Behavioural text, however the link will be replaced with a weblink to an animated video. This video has been designed through an extensive co-design process involving several behavioural change techniques designed to overcome barriers highlighted in this qualitative work.
  Behavioural Message + Video: Messaging as above. The video also includes information on emotional consequences, problem solving, anticipated regret, reducing negative emotions and credible source techniques.
Arm/Group | Usual Care- Open | Behavioural Message- Open | Behavioural Message + Video- Open
Number analyzed (Participants) | 8654 | 8095 | 8271
participants | 4104 | 3909 | 3978

5. Secondary Outcome: No. of Participants Taking up Breast Cancer Screening, Three Months After the Initial Invitation Letter, Amongst Those With Different Screening History
Description: No. of participants taking up breast cancer screening, three months after the initial invitation letter, amongst those with different screening history
Time Frame: 3 months
Population: Timed Appointment
Measure: Number; unit: participants
Arm/Group | Usual Care | Behavioural Message | Behavioural Message + Video
Number analyzed (Participants) | 3094 | 2952 | 2981
participants
  First Time Invitee: number analyzed (Participants) | 858 | 881 | 861
  First Time Invitee | 406 | 379 | 394
  Not First Time Invitee: number analyzed (Participants) | 2236 | 2071 | 2120
  Not First Time Invitee | 1820 | 1686 | 1743

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Usual Care | Behavioural Message | Behavioural Message + Video
All-Cause Mortality (participants affected / at risk) | 0/11748 | 0/11047 | 0/11252
Serious Adverse Events (participants affected / at risk) | 0/11748 | 0/11047 | 0/11252
Other Adverse Events (participants affected / at risk) | 0/11748 | 0/11047 | 0/11252

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/71/NCT05395871/Prot_SAP_000.pdf